CLINICAL TRIAL: NCT01158352
Title: Study to Evaluate the Effect of Short Treatment With Nutritional Supplementation Standardized Formula, on Growth and Weight Gain in Short and Lean Prepubertal Children
Brief Title: Study to Evaluate the Effect of Short Treatment With Nutritional Supplementation Standardized Innovative Formula, on Growth and Weight Gain in Short and Lean Prepubertal Children
Acronym: Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rmc005547ctil
Record Dates: First submitted 2010-06-27; First posted 2010-07-08 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Growth; Low Weight; Low Height
Keywords: Growth; Low weight; Low height; Nutritional Formula
MeSH Terms: conditions — Thinness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplemntation formula (Experimental): Nutritional supplementation standardized formula (powder added to liquids or food) containing 25% of recommended DRI for calories, high protein (20% of calories) and multi vitamins and mineral(25%-100% of DRI for recommended daily allowance or adequate intake)
  Interventions: Dietary Supplement: Nutritional supplementation formula
- Placebo Comparator (Placebo Comparator): Placebo low caloric formula (Powder added to liquids or food, without added vitamins and minerals
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation formula — Nutritional supplementation formula
  Arms: Nutritional supplemntation formula
Dietary Supplement: Placebo Comparator — Placebo low caloric formula (Powder added to liquids or food, without added vitamins and minerals
  Arms: Placebo Comparator

SUMMARY:
Study design:

Double blind, randomized, placebo controlled study.The proposed study will consist of two main segments:

1. Segment 1 is aimed to assess the effect of 6-12 months treatment with nutritional supplementation standardized formula, in short and lean prepubertal children on weight SDS, height SDS, BMI SDS and growth velocity
2. Segment 2 is aimed to explore the eating behavior of idiopathic short stature and lean prepubertal children against their sibling who have a normal height and body weight and to find out whether there is a difference in eating patterns and quality of life between idiopathic short stature and lean prepubertal children and children with normal height and body weight

Segment 1

Population:

200 subjects and controls will be recruited to segment 1 of the proposed study, 100 at each group.

Participants will be recruited from healthy children who will be referred to either the institute for endocrinology or the gastroenterology unit, at Schneider Children's Medical Center for growth assessment, due to low height and weight, in whom, no gastrointestinal morbidity or other underlying cause was found.

Methods:

Randomization & Blinding:

Participants will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1. Both participants and study team will be blinded to the type of treatment that each patient will receive during the first 6 months of the study.

Treatment:

Participants in the intervention group will be treated with a nutritional supplementation standardized formula.Participants in the control group will be instructed to consume the same volume of formula as was calculated if they were in the intervention group.

Treatment duration:

The study will be divided into two treatment periods: 6 months of intervention versus active placebo followed with additional 6 months (an extension period), in which participants at the intervention group will be offered to extend the intervention period and participants at the control arm will be offered to switch to the intervention group.

Study Schedule:

Follow up visits will take place at 0, 3, 6, 9 and 12 months and will include:

1. Demographic data, medical history and growth data (month 0):

   Demographic parameters, including birth date, gender, birth weight and length for gestational age, medical history and growth data, including height velocity, parent's and sibling's weight and height will be documented from patient's file.
2. Nutritional assessment
3. Anthropometric assessment (months 0, 3, 6, 9 12):

   1. Height without shoes
   2. Length
   3. Weight with light cloths and without shoes
   4. MAC
   5. Body mass index (BMI) will be calculated from children's weight and height and age and gender specific BMI SDS will be calculated
   6. Body composition assessment using the method of bioelectrical impedance
4. Laboratory parameters (months 0, 6 and 12):
5. Sleeping Questionaire

Segment 2:

86 subjects and controls will be recruited to segment 2 of the proposed study

Population:

Short and lean prepubertal children participating at segment 1 of the study and who are at study entry under 10th percentile in height, when the weight percentile is equal or smaller to the height percentile. Only participants from segment 1 who have siblings with normal height and body weight for age and gender, will be able to participate in segment 2 of the study

Control group 1:

Sibling of participants in segment 1 of the study, who have a normal height- above 25th percentile and normal BMI for age and gender- above 5th percentile and under 85th percentile.

Control group 2:

Healthy children from the community who have a normal height above 25th percentile and normal BMI for age and gender above 5th percentile and under 85th percentile

Segment 2 of the study will be designed as a case- control study and will focus on the eating patterns, sleeping patterns and quality of life of participants at segment 1 at time 0 month of the study, before the beginning of the nutrition intervention. These findings will be compared to data of a control group, which will be comprised of siblings of participants in segment 1, with normal height and body weight which are matched in age.

ELIGIBILITY:
Inclusion Criteria for participants at the intervention group (segments 1&2):

1. Girls aged 3-7 years old and boys aged 3-8 years old
2. Prepubertal - tanner stage 1
3. Height, weight and BMI < 10th percentile for age and gender
4. Availability of growth velocity data for at least 4 months prior to study entry.
5. Signing inform consent forms

Exclusion Criteria for participants at the intervention group (segments 1):

1. Diagnosis of GH Deficiency or treatment with GH
2. Any known chronic disease or dysmorphic syndrome including: bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardial, renal or pulmonary problems
3. Any known gastrointestinal problem including absorption problems
4. Any known organic reason for slow growth
5. Any chronic treatment with medication that might effects appetite (for example SSRI's), weight or Growth.

Inclusion Criteria for participants at the control group (segments 2):

1. Girls aged 3-8 years old and boys aged 3-9 years old
2. Prepubertal - tanner stage 1
3. Height ≥ 25th percentile for age and gender
4. Proper proportion between weight and height- 5th ≤ BMI ≤ 85th
5. Signing inform consent forms

Exclusion Criteria for participants at the control group (segments 2):

1. Diagnosis of GH Deficiency or treatment with GH
2. Any known chronic disease or dysmorphic syndrome including: bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardial, renal or pulmonary problems
3. Any known gastrointestinal problem including absorption problems
4. Any known organic reason for slow growth
5. Any chronic treatment with medication that might effects appetite (for example SSRI's), weight or Growth
6. Children with growth faltering during the previous year

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Height SDS (standard deviation score) | At 12 months
  standard deviation score of patient's height at 12 months

SECONDARY OUTCOMES:
Weight SDS (standard deviation score) | At 12 months
  Standard deviation score of patient's weight at 12 months
Weight/Height SDS (standard deviation score) | At 12 months
  Standard deviation score of patient's Weight / Height ratio at 12 months
BMI SDS (standard deviation score) | At 12 months
  standard deviation score of patient's BMI at 12 months
Growth Velocity | At 12 months
5.Sleeping Questionaire | At 12 months
Child Eating Behaviour Questionaire (CEBQ) | At 12 months
3-day food diary | At 12 months
Physical activity questionnaire | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schenider Children's Medical
Locations (1):
- Schneider Children's Medical center, Petaach-Tikva, Israel

REFERENCES:
- [Derived] Yackobovitch-Gavan M, Lebenthal Y, Lazar L, Shalitin S, Demol S, Tenenbaum A, Shamir R, Phillip M. Effect of Nutritional Supplementation on Growth in Short and Lean Prepubertal Children after 1 Year of Intervention. J Pediatr. 2016 Dec;179:154-159.e1. doi: 10.1016/j.jpeds.2016.08.100. Epub 2016 Sep 30. PMID 27697330
- [Derived] Lebenthal Y, Yackobovitch-Gavan M, Lazar L, Shalitin S, Tenenbaum A, Shamir R, Phillip M. Effect of a nutritional supplement on growth in short and lean prepubertal children: a prospective, randomized, double-blind, placebo-controlled study. J Pediatr. 2014 Dec;165(6):1190-1193.e1. doi: 10.1016/j.jpeds.2014.08.011. Epub 2014 Sep 17. PMID 25241181